CLINICAL TRIAL: NCT05870722
Title: Pinpointing the Factors Affecting Clinical Study Experiences of Schizophrenia Patients
Brief Title: An In Depth Study Evaluating The Experiences of Patients In Schizophrenia Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84771018
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, research participation has been biased toward certain demographics. However, there is a shortage of studies that delve into the underlying factors that influence patient participation, both positively and negatively.

Several people will be invited to enroll in this study so that it may collect a variety of data about schizophrenia clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

The data collected from this study will be analyzed and used to improve the experiences of future schizophrenia patients who are recruited for medical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with schizophrenia
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenia patients who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a schizophrenia research | 3 months
Rate of patients who remain in schizophrenia clinical trial to trial completion | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barnett PG, Scott JY, Rosenheck RA; CSP 555 Study Group. How do clinical trial participants compare to other patients with schizophrenia? Schizophr Res. 2011 Aug;130(1-3):34-9. doi: 10.1016/j.schres.2011.03.033. Epub 2011 Apr 22. PMID 21514794
- [Background] Kishimoto T, Robenzadeh A, Leucht C, Leucht S, Watanabe K, Mimura M, Borenstein M, Kane JM, Correll CU. Long-acting injectable vs oral antipsychotics for relapse prevention in schizophrenia: a meta-analysis of randomized trials. Schizophr Bull. 2014 Jan;40(1):192-213. doi: 10.1093/schbul/sbs150. Epub 2012 Dec 17. PMID 23256986
- [Background] Maric NP, Jovicic MJ, Mihaljevic M, Miljevic C. Improving Current Treatments for Schizophrenia. Drug Dev Res. 2016 Nov;77(7):357-367. doi: 10.1002/ddr.21337. Epub 2016 Sep 16. PMID 27633376

DOCUMENTS (1):
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT05870722/ICF_000.pdf